CLINICAL TRIAL: NCT01083641
Title: A Phase II Study of High Dose Estradiol in Metastatic Triple Negative Breast Cancer
Brief Title: Estrogen for Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: did not meet efficacy goals after interim analysis
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO09711; H-2009-0172 (Other: Institutional Review Board); NCI-2011-00618 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); P30CA014520 (NIH)
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2017-03

CONDITIONS: Female Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Estrogen Therapy (Experimental): Estrogen therapy
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol — 10mg oral three times daily

SUMMARY:
The purpose of this study is to determine the effectiveness of Estradiol treatment for advanced breast cancer that is hormone receptor negative and Her2/neu negative. The study will also use tumor tissue from your original diagnosis or from a biopsy you may have had for your cancer to look at hormone receptors in the lab. The tissue left over from your previous surgery or a previous biopsy will be used for research tests to check whether a different estrogen receptor (estrogen receptor beta) is seen in the tumor and if that makes estrogen work better.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed breast cancer which is metastatic.
* A formalin-fixed paraffin embedded tumor block (preferred) or unstained slides must be available from either a prior biopsy of the primary tumor or a metastatic site. .
* Primary tumor or metastatic biopsy lacking estrogen and progesterone receptor and Her2 negative
* Patients must have measurable disease.
* Eastern Cooperative Oncology Group performance status 0-1.
* Patients with bone metastasis at baseline must agree to treatment with intravenous bisphosphonates
* Subjects may have had 0-4 lines of prior systemic chemotherapy or targeted therapy regimens administered for treatment of their metastatic breast cancer.
* Age >18 years
* Life expectancy of greater than 3 months.
* Patients must have adequate organ and marrow function as defined below:

Exclusion Criteria:

* systemic chemotherapies, targeted therapies or radiotherapy for their cancer within 2 weeks prior to entering the study
* Patients receiving any other investigational agents for breast cancer treatment.
* Patients with known brain metastases are excluded 3.2.4 History of allergic reactions attributed to compounds of similar chemical or biologic composition to estradiol.
* Patients with any condition of the gastrointestinal tract that is expected to result in an inability to take oral medication
* Dysfunctional or post-menopausal vaginal bleeding.
* Uncontrolled hypercalcemia/hypocalcemia
* Prior history of or active thrombophlebitis, cerebral vascular accident, myocardial infarction, deep venous thrombosis or pulmonary embolism.
* History of or active hepatic adenoma.
* Uncontrolled intercurrent illness
* Pregnant women are excluded from this study
* Patients with bone metastasis are excluded if they are unable to receive intravenous bisphosphonate therapy due to the risk for developing hypercalcemia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari B Wisinski, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter phase 2 study was conducted through the Wisconsin Oncology Network. Subjects were recruited from February 2010 through March 2013.
Period: Overall Study
Arm/Group | Estrogen Therapy
Started | 17
Completed | 15
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Adult women with measurable advanced TNBC.
Arm/Group | Estrogen Therapy
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 57.9 [34 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 17
Stage at Diagnosis [Count of Participants; unit: Participants] — Breast cancer stages:
  I: tumor =<2cm and no lymph nodes involved.
  II: tumor measures 2cm-5cm, or cancer has spread to lymph nodes under the arm on the same side as the breast cancer.
  III: Tumor >2cm and cancer is extensive in the underarm lymph nodes, or has spread to other lymph nodes or tissues near the breast.
  IV: Cancer has spread beyond the breast, underarm, and internal mammary lymph nodes to other parts of the body near to or distant from the breast.
  Participants
    Stage I | 3
    Stage II | 9
    Stage III | 4
    Stage IV | 1

OUTCOME MEASURES:

1. Primary Outcome: Determine Tumor Objective Response (OR) Rates
Description: OR=complete response (CR) + partial response (PR) as defined by RECIST version 1.1, where CR=disappearance of all target lesions, and PR=At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 4 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Estrogen Therapy
Number analyzed (Participants) | 15
percentage of participants | 5.9 [0.2 to 28.7]

2. Secondary Outcome: Clinical Benefit (CB)
Description: Defined as complete response, partial response, or stable disease at > 16 weeks
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Estrogen Therapy
Number analyzed (Participants) | 17
Participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease at > 16 weeks | 1
  Stable Disease < 16 weeks | 2

3. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Estrogen Therapy
Number analyzed (Participants) | 17
months | 1.9 [1.3 to 4.0]

4. Secondary Outcome: Median Overall Survival (OS)
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Estrogen Therapy
Number analyzed (Participants) | 17
months | 7.6 [3.9 to 20.4]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 4 years.
Description: Toxicity evaluations including history, examination, and laboratory analysis occurred on day 1 of each cycle.
Arm/Group | Estrogen Therapy
Serious Adverse Events (participants affected / at risk) | 4/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estrogen Therapy (N=17)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Pain- back (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1)
Thrombosis/Thrombus/embolism (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estrogen Therapy (N=17)
Albumin, serum-low (hypoalbuminemia) Count (Metabolism and nutrition disorders) | 10 (11)
Alkaline phosphatase Count (Metabolism and nutrition disorders) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) Count (Metabolism and nutrition disorders) | 2 (2)
Anorexia Count (Gastrointestinal disorders) | 4 (4)
AST, SGOT(serum glutamic oxaloacetic transaminase) Count (Metabolism and nutrition disorders) | 3 (5)
Calcium, serum-low (hypocalcemia) Count (Metabolism and nutrition disorders) | 3 (4)
Confusion Count (Nervous system disorders) | 1 (1)
Constipation Count (Gastrointestinal disorders) | 4 (5)
Cough Count (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Creatinine Count (Metabolism and nutrition disorders) | 1 (1)
Dermal change lymphedema, phlebolymphedema Count (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin Count (Skin and subcutaneous tissue disorders) | 1 (2)
Diarrhea Count (Gastrointestinal disorders) | 1 (2)
Distension/bloating, abdominal Count (Gastrointestinal disorders) | 3 (3)
Dizziness Count (Nervous system disorders) | 3 (3)
Dry mouth/salivary gland (xerostomia) Count (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) Count (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Edema: limb Count (Blood and lymphatic system disorders) | 6 (7)
Fatigue (asthenia, lethargy, malaise) Count (General disorders) | 13 (23)
Glucose, serum-high (hyperglycemia) Count (Metabolism and nutrition disorders) | 3 (3)
Glucose, serum-low (hypoglycemia) Count (Metabolism and nutrition disorders) | 1 (1)
Hair loss/alopecia (scalp or body) Count (Skin and subcutaneous tissue disorders) | 1 (1)
Hemoglobin Count (Blood and lymphatic system disorders) | 6 (7)
Hemorrhage Count (Blood and lymphatic system disorders) | 5 (7)
Hypertension Count (Cardiac disorders) | 1 (1)
Infection Count (Infections and infestations) | 4 (4)
Leukocytes (total WBC) Count (Blood and lymphatic system disorders) | 3 (5)
Lymphedema-related fibrosis Count (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia Count (Blood and lymphatic system disorders) | 1 (1)
Mood alteration - Anxiety Count (Nervous system disorders) | 1 (1)
Mood alteration - Depression Count (Nervous system disorders) | 2 (2)
Nausea Count (Gastrointestinal disorders) | 11 (12)
Neuropathy: sensory Count (Nervous system disorders) | 6 (8)
Neutrophils/granulocytes (ANC/AGC) Count (Blood and lymphatic system disorders) | 1 (1)
Pain Count (General disorders) | 14 (26)
Potassium, serum-low (hypokalemia) Count (Metabolism and nutrition disorders) | 2 (4)
Pruritus/itching Count (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, __) Count (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sodium, serum-low (hyponatremia) Count (Metabolism and nutrition disorders) | 1 (1)
Vaginal discharge (non-infectious) Count (Reproductive system and breast disorders) | 4 (4)
Vision-flashing lights/floaters Count (Eye disorders) | 1 (2)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) Count (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting Count (Gastrointestinal disorders) | 5 (5)
Weight gain Count (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No